CLINICAL TRIAL: NCT03818919
Title: Traditional vs. Nonopioid Analgesia After Rotator Cuff Repair
Brief Title: Nonopioid Analgesia After Rotator Cuff Repair
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Vasilios Moutzouros, Senior Staff, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123191
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Celecoxib; Ketorolac; Acetaminophen; Gabapentin; Diazepam; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Post-Operative Non Opioid Pain Protocol (Experimental): Patients in this group will be administered a novel multimodal pain protocol post-operatively consisting of: Celecoxib, Ketorolac, Gabapentin, Acetaminophen, Diazepam
  Interventions: Drug: Celecoxib; Drug: Ketorolac; Drug: Gabapentin; Drug: Acetaminophen; Drug: Diazepam
- Post-Operative Traditional Pain Protocol (Active Comparator): Patients will be administered a traditional post-operative pain protocol consisting of: Hydrocodone-Acetaminophen Cap 5-500
  Interventions: Drug: Hydrocodone-Acetaminophen

INTERVENTIONS:
Drug: Celecoxib — Post-Operative Non Opioid Pain Protocol
  Other Names: Celebrex
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Ketorolac — Post-Operative Non Opioid Pain Protocol
  Other Names: Tylenol
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Gabapentin — Post-Operative Non Opioid Pain Protocol
  Other Names: Neurontin
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Acetaminophen — Post-Operative Non Opioid Pain Protocol
  Other Names: Tylenol
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Diazepam — Post-Operative Non Opioid Pain Protocol
  Other Names: Valium
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Hydrocodone-Acetaminophen — Traditionally used narcotic pain protocol
  Other Names: Norco
  Arms: Post-Operative Traditional Pain Protocol

SUMMARY:
This is a randomized, single blinded, standard of care controlled clinical trial. This project aims to compare postoperative pain control in patients in two treatment arms of rotator cuff repair: a treatment group given a nonopioid pain control regimen, and a standard of care control group given standard opioid pain control regimen

DETAILED DESCRIPTION:
Study Design: This is a randomized, single blinded, standard of care-controlled clinical trial. All adult patients over eighteen desiring rotator cuff repair will be eligible. Nonnarcotic postoperative pain control regimen described below were chosen based on previous studies in fracture care and joint arthroplasty.

Patients will be consented and recruited. Once participation has been determined and consent obtained, the names of participating patients will be provided to the research pharmacy. Patients will be randomized with a computer-generated table in 2 patient blocks by the research pharmacy. Patients postoperative analgesia will be divided into one of the following 2 treatment arms: 1) A novel nonopioid pain protocol or 2) traditional narcotic pain analgesia

Primary endpoints is reduction in pain as measured by visual analogue scale and Patient-Reported Outcomes Measurement Information System. The endpoints will be collected at each post-operative day using a journal. Moreover, endpoints will be collected at the patient's first post-operative appointment. These appointments are scheduled within one-week of the index procedure.

Statistical Analysis: All continuous data will be analyzed using independent 2-group t tests and reported as means ± standard deviations. Categorical data will be compared between the 2 groups using chi-square tests and reported as counts and percentages. A preliminary test to confirm the quality of variances will be conducted prior to utilizing the t test to confirm the appropriate statistical analysis. Nonparametric equivalents Wilcoxon rank-sum and Fisher exact tests will be used as needed for nonnormal distributions and low variable numbers, respectively. A multivariable regression analysis was performed to assess for potential confounding demographic variables.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over age 18 and scheduled for a primary or revision rotator cuff repair

Exclusion Criteria:

* Exclusion criteria will include patients with a medical history of known allergies or intolerance to allergies or intolerance to Celebrex, Tylenol, Neurontin, dexamethasone, tramadol, substantial alcohol or drug abuse, and pregnancy, history of narcotics within 6 months of surgery, renal impairment, peptic ulcer disease, GI bleeding. Secondary exclusion criterion is an intact rotator cuff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toufic R Jildeh, MD, Principal Investigator — Resident
Locations (1):
- Health Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Per Request

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post-Operative Non Opioid Pain Protocol | Post-Operative Traditional Pain Protocol
Started | 35 | 35
Completed | 17 | 23
Not Completed | 18 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-Operative Non Opioid Pain Protocol | Post-Operative Traditional Pain Protocol | Total
Number analyzed (Participants) | 17 | 23 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 20 | 36
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.1) | 55.9 (7.2) | 54.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 9 | 13 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 7 | 14 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
BMI [Mean (Standard Deviation); unit: kg/m2] | 32.2 (6.8) | 29.9 (5.5) | 30.8 (5.7)
Preoperative block [Count of Participants; unit: Participants]
  Supraclavicular | 3 | 5 | 8
  Interscalene | 14 | 18 | 32
Tear size [Count of Participants; unit: Participants]
  less than 1 cm | 1 | 4 | 5
  1-3cm | 11 | 16 | 27
  3-5cm | 5 | 2 | 7
  greater than 5cm | 0 | 1 | 1
Tendons involved in surgery [Mean (Standard Deviation); unit: number of tendons involved] | 1.7 (0.4) | 1.4 (0.8) | 1.55 (0.6)
Concomitant procedures [Count of Participants; unit: Participants]
  None | 0 | 2 | 2
  Biceps Tenotomy | 2 | 2 | 4
  Biceps Tenodesis | 4 | 3 | 7
  DCE | 1 | 2 | 3
  SAD | 10 | 14 | 24
Anchors used in Surgery [Mean (Standard Deviation); unit: number of anchors used] | 2.7 (0.8) | 2.6 (1.1) | 2.6 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Pain Levels
Description: Patients record pain levels using Visual analog scales for 10 days post-operatively. The visual analog scale ranges from 0 (no pain) to 10 (worst pain). Average daily pain was calculated for each patient. Higher values portend worse control.
Time Frame: day 10 post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post-Operative Non Opioid Pain Protocol | Post-Operative Traditional Pain Protocol
Number analyzed (Participants) | 17 | 23
units on a scale | 2.4 (2.1) | 3 (1.8)

2. Primary Outcome: Patient-Reported Outcomes Measurement Information System
Description: Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS PI) for 10 days post-operatively. PROMIS-PI scale ranges from 0 (no pain interference ) to 100 (most pain interference). Average PROMIS PI values were calculated. A higher score indicates more pain interference.
Time Frame: day 10 post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post-Operative Non Opioid Pain Protocol | Post-Operative Traditional Pain Protocol
Number analyzed (Participants) | 17 | 23
units on a scale | 59.3 (8.5) | 60.0 (9.3)

ADVERSE EVENTS:
Time Frame: 10 days postop
Arm/Group | Post-Operative Non Opioid Pain Protocol | Post-Operative Traditional Pain Protocol
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/23
Other Adverse Events (participants affected / at risk) | 8/17 | 10/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Post-Operative Non Opioid Pain Protocol (N=17) | Post-Operative Traditional Pain Protocol (N=23)
GI adverse effects (Gastrointestinal disorders) | 8 | 10 — includes constipation, diarrhea, nausea, and upset stomach

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT03818919/Prot_SAP_001.pdf